CLINICAL TRIAL: NCT02964780
Title: Study on Mechanisms of Changes in Liver Disease and Sex Steroid Metabolism During Weight Loss
Acronym: SMELSS
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201526667
Record Dates: First submitted 2016-10-24; First posted 2016-11-16 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Gastric Bypass Surgery: Solid mixed meal tolerance test, MRI, CT, anthropometrics, liver biopsies, fat biopsies, muscle biopsies
  Interventions: Procedure: Gastric bypass surgery
- Conservative weight loss: Solid mixed meal tolerance test, MRI, CT, anthropometrics, liver biopsies, fat biopsies, muscle biopsies
  Interventions: Behavioral: Conservative weight loss program

INTERVENTIONS:
Procedure: Gastric bypass surgery
  Groups: Gastric Bypass Surgery
Behavioral: Conservative weight loss program
  Groups: Conservative weight loss

SUMMARY:
The main objective of the study is to gain insight in the early dynamics and mechanisms of recovery of liver disease and sex steroid metabolism during weight loss in obese men and women and to investigate whether surgical weight loss has differential effects as compared to weight loss with life style measures. In addition, we want to evaluate the postprandial hypoglycemic reactive syndrome (PPHRS) in these patients using a standard chewable meal.

Secondary objectives are investigating determinants for the changes in sex steroids, liver disease and PPHRS. Possible determinants to be investigated are adipocytokine secretion patterns, body composition, resting metabolism rate, weight loss per se and changes in fat distribution, parameters of fatty acid metabolism, … .

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* BMI > 35 kg/m²

Exclusion Criteria:

* Primary or secondary hypogonadism due to genetic causes (Kallman syndrome etc.), tumors, infiltrative diseases, infections, pituitary apoplexy, trauma, critical illness, chronic systemic illness or intentional.
* Type 2 Diabetes Mellitus treated with insulin or GLP-1 analogues
* Current or recent use of insulin, corticosteroids, opiates (on a daily basis), growth hormones, androgen- or estrogen analogs, levothyroxine, anti-retroviral drugs or antipsychotics
* Cancer (within < 5 years)
* High-grade malignancies
* Serious co-morbidities such as renal, hepatic of cardiac failure
* Known or suspected abuse of alcohol or narcotics
* Mental incapacity, unwillingness, or language barrier precluding adequate understanding or cooperation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obesity class 3 who want to reduce weight
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sex steroids | Baseline, 3 weeks, 6 weeks, 6 months, 1 year.
  The change in sex steroids will be compared between the conservative and the gastric bypass group.
Change from baseline in liver fat | Baseline, 6 months, 1 year
  The change in liver steatose will be compared between the conservative and the gastric bypass group
Correlation in changes in liver fat en changes in sex steroids | baseline, 6 months, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology, UZ Ghent Hospital, Ghent, Belgium